CLINICAL TRIAL: NCT05152823
Title: Phase I/IIa Intrathecal Gene Delivery Clinical Trial for IGHMBP2-Related Diseases
Brief Title: Gene Therapy for IGHMBP2-Related Diseases
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Megan Waldrop (Other)
Responsible Party: Sponsor-Investigator, Megan Waldrop, Professor of Neurology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002143
Record Dates: First submitted 2021-11-25; First posted 2021-12-10 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: SMARD1; CMT2S
Keywords: IGHMBP2
MeSH Terms: conditions — Spinal muscular atrophy with respiratory distress 1 | interventions — Genetic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Intrathecal Delivery (Experimental)
  Interventions: Biological: Gene Therapy

INTERVENTIONS:
Biological: Gene Therapy — AAV9 carrying the IGHMBP2 gene.

SUMMARY:
Open-label, single intrathecal injection study of a AAV9 vector carrying the IGHMBP2 gene for IGHMBP2-related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of two pathogenic variants in the IGHMBP2 gene from a CLIA-certified lab
* Pre-ambulant (not yet walking and less than 18 months) or ambulant (as defined by the ability to walk 10 meters without assistance) or non-ambulant (inability to walk more than 10 meters unassisted)
* Ability to cooperate with functional assessments as per PI's discretion

Exclusion Criteria:

* Prior participation in a gene or cell therapy program for any kind.
* Immunizations of any kind in the month prior to the study.
* Active infection based on clinical observations
* Serological evidence of HIV infection, or Hepatitis B or C infection
* Diagnosis of (or ongoing treatment for) an autoimmune disease
* Persistent leukopenia or leukocytosis (WBC ≤ 3.5 10^3/μL or ≥ 20.0 10^3/μL) or an absolute neutrophil count < 1.5 10^3/μL
* Abnormal liver function as indicated by an elevated GGT (>2X normal if no other laboratory abnormalities), bilirubin and/or abnormal PT/INR
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer
* AAV9 binding antibody titers > 1:50 as determined by ELISA immunoassay performed by Athena Diagnostics
* Abnormal laboratory values in the clinically significant range, based upon normal values in the Nationwide Children's Hospital Laboratory
* Diagnosis of any other systemic illness that increases the risk of gene transfer per the PI's opinion; Has a medical condition or extenuating circumstance that, in the opinion of the PI, might compromise the subject's ability to comply with the protocol required testing or procedures or compromise the subject's well-being, safety, or clinical interpretability
* Any requirement for immune modulatory therapy and for which it would be unsafe for the subject to undergo an appropriate wash out period
* Contraindication for intrathecal injection
* A positive JCV antibody test of >0.40

Ages: 2 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Monitoring for the development of unacceptable toxicity. | 3 years
  Unacceptable toxicity is defined as the occurrence of two or more unexpected Grade III or higher treatment-related toxicities, as defined by CTCAE 5.0.

SECONDARY OUTCOMES:
For pre-ambulant participants, ages less than 18 months, change in the Neuromuscular Gross Motor Outcome (GRO) from baseline | Days 90 and 180, Months 12, 18, 24 and 36
For ambulant participants, change in the 100-meter timed test from baseline | Days 90 and 180, Months 12, 18, 24 and 36
For non-ambulant participants, ages 18 months to 6 years, change in the Neuromuscular Gross Motor Outcome (GRO) from baseline | Days 90 and 180, Months 12, 18, 24 and 36
For non-ambulant participants, ages greater than 6 years, change in the revised upper limb module for SMA (RULM) from baseline | Days 90 and 180, Months 12, 18, 24 and 36

CONTACTS AND LOCATIONS:
Overall Officials: Megan Waldrop, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Grohmann K, Schuelke M, Diers A, Hoffmann K, Lucke B, Adams C, Bertini E, Leonhardt-Horti H, Muntoni F, Ouvrier R, Pfeufer A, Rossi R, Van Maldergem L, Wilmshurst JM, Wienker TF, Sendtner M, Rudnik-Schoneborn S, Zerres K, Hubner C. Mutations in the gene encoding immunoglobulin mu-binding protein 2 cause spinal muscular atrophy with respiratory distress type 1. Nat Genet. 2001 Sep;29(1):75-7. doi: 10.1038/ng703. PMID 11528396
- [Background] Saladini M, Nizzardo M, Govoni A, Taiana M, Bresolin N, Comi GP, Corti S. Spinal muscular atrophy with respiratory distress type 1: Clinical phenotypes, molecular pathogenesis and therapeutic insights. J Cell Mol Med. 2020 Jan;24(2):1169-1178. doi: 10.1111/jcmm.14874. Epub 2019 Dec 4. PMID 31802621
- [Background] Guenther UP, Handoko L, Varon R, Stephani U, Tsao CY, Mendell JR, Lutzkendorf S, Hubner C, von Au K, Jablonka S, Dittmar G, Heinemann U, Schuetz A, Schuelke M. Clinical variability in distal spinal muscular atrophy type 1 (DSMA1): determination of steady-state IGHMBP2 protein levels in five patients with infantile and juvenile disease. J Mol Med (Berl). 2009 Jan;87(1):31-41. doi: 10.1007/s00109-008-0402-7. Epub 2008 Sep 18. PMID 18802676
- [Background] Viguier A, Lauwers-Cances V, Cintas P, Manel V, Peudenier S, Desguerre I, Quijano-Roy S, Vanhulle C, Fradin M, Isapof A, Jokic M, Mathieu-Dramard M, Dieterich K, Petit F, Magdelaine C, Giuliano F, Gras D, Haye D, Nizon M, Magen M, Bieth E, Cances C. Spinal muscular atrophy with respiratory distress type 1: A multicenter retrospective study. Neuromuscul Disord. 2019 Feb;29(2):114-126. doi: 10.1016/j.nmd.2018.10.002. Epub 2018 Oct 31. PMID 30598237
- [Background] Tomaselli PJ, Horga A, Rossor AM, Jaunmuktane Z, Cortese A, Blake JC, Zarate-Lopez N, Houlden H, Reilly MM. IGHMBP2 mutation associated with organ-specific autonomic dysfunction. Neuromuscul Disord. 2018 Dec;28(12):1012-1015. doi: 10.1016/j.nmd.2018.08.010. Epub 2018 Aug 29. PMID 30385095
- [Background] Eckart M, Guenther UP, Idkowiak J, Varon R, Grolle B, Boffi P, Van Maldergem L, Hubner C, Schuelke M, von Au K. The natural course of infantile spinal muscular atrophy with respiratory distress type 1 (SMARD1). Pediatrics. 2012 Jan;129(1):e148-56. doi: 10.1542/peds.2011-0544. Epub 2011 Dec 12. PMID 22157136
- [Background] Cottenie E, Kochanski A, Jordanova A, Bansagi B, Zimon M, Horga A, Jaunmuktane Z, Saveri P, Rasic VM, Baets J, Bartsakoulia M, Ploski R, Teterycz P, Nikolic M, Quinlivan R, Laura M, Sweeney MG, Taroni F, Lunn MP, Moroni I, Gonzalez M, Hanna MG, Bettencourt C, Chabrol E, Franke A, von Au K, Schilhabel M, Kabzinska D, Hausmanowa-Petrusewicz I, Brandner S, Lim SC, Song H, Choi BO, Horvath R, Chung KW, Zuchner S, Pareyson D, Harms M, Reilly MM, Houlden H. Truncating and missense mutations in IGHMBP2 cause Charcot-Marie Tooth disease type 2. Am J Hum Genet. 2014 Nov 6;95(5):590-601. doi: 10.1016/j.ajhg.2014.10.002. Epub 2014 Oct 30. PMID 25439726